# Statistical Analysis Plan

Protocol Number: MT-186-J20

# Dose Finding Study of MCI-186 in Acute Ischemic Stroke

Version Number: 02.00

Date: 19 July, 2018

NCT number: NCT03346538

Protocol No. MCI-186-J20

Date: 19 July, 2018

# STATISTICAL ANALYSIS PLAN

Protocol No.

MCI-186-J20

Protocol Title

Dose Finding Study of MCI-186 in Acute Ischemic Stroke

Version History

Version 01.00 First approved version / 17 July, 2018

Version 02.00 First approved version / 19 July, 2018

Author

Protocol No: MCI-186-J20

Version 02.00

Author:

Date: 19 July, 2018

Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation Protocol No. MCI-186-J20 Date: 19 July, 2018

# Statistical Analysis Plan

Protocol Reference Number: MCI-186-J20

Dose Finding Study of MCI-186 in Acute Ischemic Stroke

PREPARED BY: Mitsubishi Tanabe Pharma Corporation

**VERSION:** 

02.00

DATE:

19 July, 2018

Author:

Date: 19 July, 2018

MCI-186-J20

Protocol No.

Protocol No. MCI-186-J20 Date: 19 July, 2018

# APPROVAL FORM

# STATISTICAL ANALYSIS PLAN

| Protocol Title | Dose Finding Stud | ly of MCI-186 in | Acute Ischemic | Stroke |
|---|---|---|---|---|
| Version | 02.00 | | | |
| Author(s) | | | | |
| Position | Biostatistics Group<br>Ikuyaku. Integrate | | | |
| Signature | | | | |
| Date | | | | |
| | on the planned analysi | | | ed the Statistical Analysis Planting. |
| MTPC Statistics | Reviewer | | | |
| Name: | Date | »: | Signature: _ | |
| Position:<br>Responsible ST | AT | | - | |
| APPROVED BY | <b>′:</b> | | | |
| MTPC Statistics | Approver : | | | |
| Name: | Date | <b>:</b> | Signature: | |
| Position:<br>Head of Regiona | al STAT | | | |
| Protocol No: MCI-186 | -J20 Versio | on 02.00 | Author: | Date: 19 July, 2018 |

Protocol No. MCI-186-J20 Date: 19 July, 2018

# TABLE OF CONTENTS

| 1. | INTRODUCTION |
|---|---|
| 2. | STUDY OBJECTIVE(S) AND ENDPOINTS 1 2.1 Study Objective(s) 1 2.2 Primary Efficacy/Safety Endpoint(s)/Assessments 1 2.3 Secondary Efficacy/Safety Endpoint(s)/Assessments 1 2.4 Safety Assessment(s) 2 2.5 Pharmacokinetics Endpoint(s)/Evaluation(s) 2 2.6 Pharmacodynamics Endpoint(s)/Evaluation(s) 2 2.7 Other Endpoint(s)/Evaluation(s) 2 |
| 3. | STUDY DESIGN |
| 4. | 4.1 Data Monitoring Board (DSMB) 7 4.2 Interim Analysis 7 |
| 5 | 4.3 Final Analysis |
| 3. | · <b>,</b> |
| 6. | GENERAL CONSIDERATIONS8 |
| 7. | STATISTICAL METHODOLOGY 9 7.1 Study Patients 9 7.1.1 Disposition of Subjects 9 7.1.2 Demographic and Other Baseline Characteristics 9 7.1.3 Medical History 10 7.1.4 Concomitant Medications and Concomitant Therapys 10 7.1.5 Study Medication Exposure 10 7.1.6 Compliance 10 |
| | 7.2 Efficacy Assessment 11 7.2.2 Primary Efficacy Endpoint 12 7.2.3 Secondary Efficacy Endpoints 12 7.2.4 Other Efficacy 13 7.2.5 Quality of Life Assessments 13 7.2.6 Exploratory endpoint 14 |
| | 7.3 Safety Assessments |

# Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation

Protocol No. MCI-186-J20 Date: 19 July, 2018

| | 7.3.3 | Vital Signs | 15 |
|----|--------------|----------------------------------------|----|
| | 7.3.4 | 12-lead ECG | 15 |
| | 7.3.5 | Physical Examinations | 16 |
| | 7.3.6 | Other Safety Assessments | 16 |
| 8. | CHANGES | FROM THE PROTOCOL | 16 |
| 9. | DATA NOT | SUMMARISED OR PRESENTED | 16 |
| 10 | . REFERENC | CES | 17 |
| 11 | . VALIDATI | ONS | 17 |
| 12 | . PROGRAM | MING AND DATA PRESENTATION CONVENTIONS | 18 |
| 13 | . LIST OF LI | STINGS, TABLES AND FIGURES | 20 |
| 14 | APPENDIX | 1 – ANALYSIS TIME WINDOW | 22 |

Version 02.00

Protocol No. MCI-186-J20 Date: 19 July, 2018

#### **ABBREVIATIONS**

#### UPDATE THE LIST AS APPROPRIATE

AE : adverse event
BI : Barthel Index
CRF : case report form
DP : decimal places
ECG : electrocardiogram

eCRF : electronic case report form

FAS : full analysis set

FIM: Functional Independence Measure

IAO : international agreed order

IMP : investigational medicinal product

MedDRA : medical dictionary for regulatory activites

mRS : modified Rankin Scale

NIHSS : National Institutes of Health Stroke Scale

PT : preferred term QC : quality control

SAP : statistical analysis plan
SAE : serious adverse event
SAF : safety population
SD : standard deviation
SOC : system organ class

TEAE : treatment emergent adverse event

WHO : World Health Organisation

Author: Date: 19 July, 2018

#### 1. INTRODUCTION

This statistical analysis plan (SAP) is based on the final protocol version 01.01 dated 1 August 2017. The plan covers statistical analysis, tabulations and listings of efficacy and safety data to investigate the efficacy and safety of MCI-186 (bolus followed by 72-hour continuous infusion) in acute ischemic stroke patients through a double-blind, parallel-group comparison with the existing MCI-186 dosing regimen as the control.

The SAP is prepared by Mitsubishi Tanabe Pharma Corporation(MTPC), Data Science Department. The statistical analyses and production of the outputs described in the SAP will be conducted and QC checked by Medical Development Business Department2 SAS Consulting Group, using SAS® 9.3 or later Software. The final analyses and outputs will be approved by Mitsubishi Tanabe Pharma Corporation, Data Science Department.

MTPC has early decided to stop subjects's recruitment based on internal decision. Therefore, the planned sample size will not be completed so that this plan will be executed based on a limited available sample size. The finding for this statistical analysis will lead to exploratory results.

#### 2. STUDY OBJECTIVE(S) AND ENDPOINTS

#### 2.1 Study Objective(s)

To investigate the efficacy and safety of MCI-186 (bolus followed by 72-hour continuous infusion) in acute ischemic stroke patients through a double-blind, parallel-group comparison with the existing MCI-186 dosing regimen as the control.

#### 2.2 Primary Efficacy/Safety Endpoint(s)/Assessments

• Primary endpoint

NIHSS (change over the 7 days from onset)

#### 2.3 Secondary Efficacy/Safety Endpoint(s)/Assessments

- Secondary endpoints
- (1) NIHSS (Day 4, Day 7, Day 10, Day 14, after 3 weeks, at discharge, after 3 months)
- (2) mRS (after 3 weeks, at discharge, after 3 months)
- (3) BI (Day 14, after 3 weeks, at discharge, after 3 months)
- (4) FIM (after 3 weeks, at discharge, after 3 months)
- (5) Start of rehabilitation

- Duration of hospitalization (6)
- Cranial imaging diagnosis (7)

#### Safety Assessment(s) 2.4

- Safety endpoints
- (1) Adverse events and adverse reactions
- (2) Neurological testsassessments
- (3) Common clinical laboratory tests
- (4) Vital signs
- (5) Standard 12-lead ECG

#### 2.5 Pharmacokinetics Endpoint(s)/Evaluation(s)

Not applicable in the study.

#### Pharmacodynamics Endpoint(s)/Evaluation(s) 2.6

Not applicable in the study.

#### Other Endpoint(s)/Evaluation(s) 2.7

Exploratory endpoint

#### STUDY DESIGN 3.

#### 3.1 **Study Design**

Phase of study: Phase 2

Study type

: Confirmatory study (planned)

Multicenter, randomized, double-blind, parallel-group study with the approved dosing regimen as the control

Date: 19 July, 2018 Version 02.00 Author: Protocol No: MCI-186-J20



#### Rationale

This study was designed as a parallel-group comparative study with the existing dosing regimen as the control in order to objectively investigate the efficacy and safety of the 72-hour continuous infusion dosing regimen. In addition, in order to minimize rater bias, a double-dummy method will be used to administer the investigational product, and the study will be conducted using a randomized, double-blind method.

#### 3.2 **Schedule of Study Procedures**

Study assessments are summarized in the Time and events schedule (Table 1).

Date: 19 July, 2018 Author:

Table 1: Assessment and Observation Schedule

| Table 1: Ass | | | | <b>Jbserv</b> | ation/ | Sched | ule | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | fore Trea | \n | | Study Drug Treatment Period | | | | | | | Observation period | | |
| Assessment<br>Time Point | Consent | Confirm ation of suitabili | Registration | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 7 | Day<br>10 | Day 14<br>or study drug<br>treatment<br>period<br>discontinuati<br>on <sup>a</sup> | After 3<br>weeks <sup>b</sup> | At<br>discharge | After 3<br>months <sup>c</sup><br>or at<br>observatio<br>n period<br>discontinu<br>ation |
| Allowable<br>Range | | | | | | | | | ±1<br>day | ±1<br>day | +1 day | ±2 days | −1 day | ±8 days<br>(+8 days) |
| Consent<br>acquisition | • | | | | | | | | | | | | | |
| Subject<br>background | | • | | | | | | | | | | | | |
| Registration/a<br>llocation | | | • | | | | | | | | | | | |
| Study drug<br>treatment | | | | <b>₹</b> 72 | -hour co | ntinuou | s infusio | 1 | <b>-</b> | | | | | |
| | Ц | | | 4- | | | Twice a c | lay for 1 | 4 days <sup>d</sup> | | | <u></u> | | |
| NIHSS | | • | | Asses | | | ed every<br>ent initia | | 7 days | • | • | • | • | • |
| mRS° | | ●f | | | | = | | | | | | • | • | • |
| BI | Ц | | | | | _ | | | | | • | • | • | • |
| FIM | Ц | | | | | | | | | | | • | • | • |
| | Ц | Div | | | | | | | | | • | • | • | • |
| Diagnostic<br>imaging | | DWI<br>T2*WI<br>FLAIR<br>MRA | | | | | DWI <sup>g</sup><br>T2*WI <sup>g</sup> | | | | DWI<br>T2*WI | | | FLAIR |
| Neurological assessments | | | | | <b>●</b> <sup>h</sup> | | | | | | • | • | • | • |
| Standard 12-<br>lead ECG | | • | | <b></b> | | | ● <sup>i</sup> | | | | | ! | | |
| Vital signs Clinical laboratory tests | | • | | | | • | ●i<br>●i | | • | | • | | | |
| (centralized<br>measurements | | | | | | | | | | | - | | | |
| Clinical<br>laboratory<br>tests (site<br>measurements | | <b>⊕</b> j | | <b>◆</b><br>Meas | | ery day | for 5 days<br>tiation <sup>k</sup> | after | | | · | | | |
| PGx blood<br>sample<br>collection | | | (Blood samples will be collected during the study from subjects who have consented to having blood samples collected for genetic analysis) | | | | | | | | | | | |
| Adverse events | | | | <b>←</b> | | | | | | | | | | |
| Concomitant medications | | | | | | | | | | | | | | |

a) If the study is discontinued during the study drug treatment period, the tests that are stipulated should be conducted at study drug treatment period discontinuation will be conducted, and whenever possible subject safety will be evaluated at 3 months after onset.

d) Twice a day, at morning and at night, for 14 days. As a rule, the drug is administered for 14 days. However, in the period after the treatment has been administered for 7 days following treatment initiation and the NIHSS assessments have been completed, treatment may be stopped only if the (sub)investigator determines that the neurological symptoms associated with the primary disease have returned to their baseline levels, the patient's condition has stabilized, and that consequently continuing to administer the study drug would not be clinically meaningful, and administering the drug would only be detrimental for the subject in that it would restrict the

b) In this study, "after 3 weeks" is defined at Day 22. If a subject is discharged within 3 weeks after treatment initiation, then the tests that are stipulated should be performed at discharge will be performed, and the tests that are scheduled for after 3 weeks will not be necessary.

In this study, after 3 months is defined as Day 85. If the study is going to be discontinued during the observation period, then the tests that are stipulated should be conducted at observation period discontinuation will be conducted, and subject safety will be assessed after 3 months whenever possible.

subject's freedom. (the subject may not be discharged).

The mRS assessments will be performed using the Japanese-language version of the mRS questionnaire (Cerebrovasc Dis 2006;21:271-278) (Attachment 2: mRS Questionnaire; Attachment 3: mRS Assessment Criteria).

The mRS assessment will also be performed prior to treatment initiation. e)

Imaging will be performed after the end of the 72-hour continuous infusion (+ 2 days).

g) h) The neurological assessments will be performed once in the period between the time of consent acquisition and Day 5.

- The standard 12-lead ECG, vital signs, and clinical laboratory tests (centralized measurements) will be performed before the end of the 72-hour continuous infusion (-1 day).
- The following tests will be conducted urgently at the hospital to confirm the patient's eligibility: WBC, RBC, hematocrit, hemoglobin, platelets, AST (GOT), ALT (GPT), LDH, ALP, γ-GTP, total bilirubin (T-Bil), CK (CPK), urea nitrogen (BUN), serum creatinine (Cre), j)
- The red blood cell (RBC), platelet (Plt), AST (GOT), ALT (GPT), LDH, ALP, total bilirubin (T-Bil), CK (CPK), urea nitrogen (BUN), k) and serum creatinine (Cre) levels only will be performed at the site every day from the day after treatment initiation through Day 5 after treatment initiation to confirm subject safety.

Version 02.00 Author: Date: 19 July, 2018 Protocol No: MCI-186-J20

# 3.3 Sample Size and Power Considerations

• A total of 336 subjects as randomized subjects

☐ Group H: 120 subjects

☐ Group L: 96 subjects

☐ Control group: 120 subjects

#### Rationale



#### 4. PLANNED ANALYSES

#### 4.1 Data Monitoring Board (DSMB)

No DSMB will be performed for this study.

#### 4.2 Interim Analysis

No interim analysis will be performed for this study.

#### 4.3 Final Analysis

All final, planned analyses identified in this SAP will be performed by MTPC Authorization of this Statistical Analysis Plan, Database Lock, Authorization of Analysis Populations and Unblinding of Treatment.

Final analysis will be done after database lock as per this SAP.

The final database lock will occur when all outstanding data queries have been resolved and the database is fully cleaned. These data will then be used to produce a full set of unblinded tables, figures and listings planned in this SAP for the Clinical Study Report. The tables, figures and listings will then be communicated to the wider study team.

#### 5. ANALYSIS POPULATION(S)

The definitions of the analysis sets are provided below. Efficacy analysis will be performed in the full analysis set (FAS) and safety analysis will be performed in the safety analysis set(SAF).

| Full<br>Analysis | FAS will be defined as all randomized subjects except for the following subjects: |
|---|---|
| Set (FAS) | - Subjects who were not with cerebral infarction |
| | - Subjects to whom the investigational product was not administered at all |
| | - Subjects for whom no post-randomization efficacy data are available |
| Safety<br>Analysis<br>Set (SAF) | The safety analysis population will be defined as all randomized subjects except for the following subjects: |
| | - All subjects to whom the investigational product was not administered a all |
| | - All subjects for whom no post-randomization safety data are available |

The acceptance or rejection of each analysis population will be treated based on the results of the data review meeting on 18 July, M200201 and M203001 are excluded from FAS and SAF.

#### 6. **GENERAL CONSIDERATIONS**

Efficacy endpoints will be analysed on the FAS population and listed on the FAS population. Subjects will be analysed according to the treatment group they were randomised to. Safety analyses will be performed on the SAF. Subjects will be analysed according to the treatment group they were actually received.

In general, continuous variables will be summarized descriptively using the number of observations (n), mean, standard deviation (SD), median, minimum and maximum. Categorical variables will be summarized using frequency counts and percentages. The denominator for the percentages will be the total number of subjects in the relevant group and population (analysis set) being presented, unless otherwise specified (e.g., on some occasions, percentages maybe calculated out of the total number of subjects with available data at a particular visit and/or time point).

For each section, baseline is the last valid assessment prior to the start of IMP administration. For numerical variables, change from baseline will be calculated as the post-baseline value minus the baseline value. If baseline value cannot be determined for a particular variable, change from baseline will not be calculated.

Data will be handled as follows.

#### (1)Definition of missing data

When test values are missing, or could not be measured because of, for example, a problem with the test sample, these values will be handled as missing. In addition, no imputation will be made in case of missing values.

#### (2) Handling of the data at measurement time points

When summarizing the data at each measurement time point, data within the analysis time windows defined in Appendix 1 will be used. If multiple values were obtained within the time window, then the value closest to the planned assessment day will be used.

Unscheduled visits will not be displayed in by-visit summary tables, but will be included in the data listings.

Listings will include scheduled, unscheduled, retest and early discontinuation data.

The date and times of start and end of IMP administration will be taken from the Electronic Case Report Form (eCRF) Dosing form.

All medical history and adverse events will be coded from the actual term using the Medical Dictionary for Regulatory Activities (MedDRA) version 20.0.

All prior and concomitant medications will be coded using the World Health Organization (WHO) drug dictionary (Version: WHO DDE B2 Mar 2017).

#### 7. STATISTICAL METHODOLOGY

#### 7.1 Study Patients

#### 7.1.1 Disposition of Subjects

Disposition of subjects will be listed.

Number and percent of subjects completed protocol scheduled visits will be presented for each study period (Study drug treatment period and Observation period). Subjects who discontinued in study drug treatment period will be summarized by reasons for discontinuation.

Number and percent of all subjects, and in each protocol defined analysis population will be presented by treatment group and overall wherever applicable.

#### 7.1.2 Demographic and Other Baseline Characteristics

Major demographic and other baseline characteristics will be listed for all subjects.

| Table2. | Variables related | to den | nographic and | l other | baseline c | haracteristics |
|---|---|---|---|---|---|---|

| Category | Variable | Data format |
|------------|--------------------------------------|-------------|
| Subject | Sex (male, female) | Binary |
| background | Age at consent acquisition (years) | Metric |
| | Weight (kg) | Metric |
| | Time from onset to first dose | Metric |
| | Pre-administration NIHSS Total Score | Metric |
| , | Spasm | Binary |
| | Race | Category |
| | Disease type | Category |
| | Japan Coma Scale | Category |
| | Medical history | Binary |
| | Concomitant Medications | Binary |
| | Concomitant Therapy | Binary |
| | Person signed Informed Consent | Category |

The above demographic and baseline data will be summarized by treatment group. Baseline Weight is taken from the assessments at the Screening visit. Age in years is derived birth date in the eCRF.

Demographic data and other baseline characteristics will be summarised for the SAF by treatment group and overall. The following demographic and other baseline characteristics will be reported for this study: Age, Sex, Weight, Time from onset to first dose, Pre-administration NIHSS Total Score, Spasm, Race, Disease type, Japan Coma Scale, Medical history, Concomitant Medications, Concomitant Therapy, Person signed Informed Consent.

#### 7.1.3 **Medical History**

All medical history data will be listed.

The frequency and percentage of subjects will be summarised by treatment group and overall for all subjects using Preferred Term nested within System Organ Class (SOC). The summary will be sorted by International Agreed Order (IAO) for SOC and alphabetical order for PT.

If Month and/or Day of medical history start date is missing, January and/or 1 will be used. If Month and/or Day of medical history end date is missing, December and/or 31 will be used.

#### 7.1.4 **Concomitant Medications and Concomitant Therapys**

All medication/therapy data will be listed.

Concomitant medications/therapys is any medications/therapys that is on-going at the time of the first dose or started after the onset of cerebral infraction. Concomitant medications/thepapys with an incomplete start date but that are still ongoing at the end of the study will be considered as concomitant medications/therapys.

#### 7.1.5 **Study Medication Exposure**

All exposure data will be listed.

The number of subjects with at least one dose of exposure of IMP will be summarised by treatment group and overall.

The duration of exposure in days will be calculated as:

1) In the case of IMP Exposure for Continuous infusion dosing regimen(hours)

Actual dosing hours =

(Date and time of last bolus dose - Date and time of first bolus dose) + sum of (Date and time of last div dose – Date and time of first div dose)

2) In the case of IMP Exposure for Approved dosing regimen(days)

Actual dosing days = Date of last dose - Date of first dose +1

If either the date of last dose or the date of first dose cannot be determined then the duration calculation will not be done. The duration of exposure will be summarised by treatment group and overall.

#### 7.1.6 Compliance

All compliance data will be summarised.

The compliance will be calculated as:

Date: 19 July, 2018 Version 02 00

- In the cese of IMP Exposure for Continuous infusion dosing regimen
   Actual dosing hours / 72 hours × 100
- 2) In the case of IMP Exposure for Approved dosing regimen

Actual dosing days / 14 days or 15 days  $\times$  100,

where if first dose is evening, then the denominater will be 15 days. Others are 14 days.

#### 7.2 .Efficacy Assessment

#### 7.2.1.1 Adjustment for Covariates

Ajustment for covariates will not be performed.

#### 7.2.1.2 Handling of Dropouts or Missing Data

Unless otherwise specified, data will be used to their maximum possible extent, but without any imputations for missing data, i.e. missing values will not be replaced or estimated.

# 7.2.1.3 Interim Analyses and Data Monitoring

No interim analysis will be performed for this study and therefore no adjustment on type 1 error will be made.

#### 7.2.1.4 Multicentre Studies

Due to the low number of subjects by centre, a centre effect was not included in any of the statistical analyses.

#### 7.2.1.5 Multiple/Comparisons/Multiplicity

The study is not powered to address multiple statistical comparisons; therefore no adjustment for multiplicity will be made.

#### 7.2.1.6 Use of an 'Efficacy Subset' of Patients

Not applicable in this study.

#### 7.2.1.7 Active-Control Studies Intended to show equivalence

Not applicable in this study.

#### 7.2.1.8 Examinations of Subgroups

Not applicable in this study.

#### 7.2.2 Primary Efficacy Endpoint

NIHSS (change over the 7 days from onset)

NIHSS value and changes from baseline will be summarized descriptively by treatment group and analysis visit.

#### 7.2.3 Secondary Efficacy Endpoints

- (1) NIHSS (Day 4, Day 7, Day 10, Day 14, after 3 weeks, at discharge, after 3 months)
- (2) mRS (after 3 weeks, at discharge, after 3 months)
- (3) BI (Day 14, after 3 weeks, at discharge, after 3 months)
- (4) FIM (after 3 weeks, at discharge, after 3 months)
- (5) Start of rehabilitation
- (6) Duration of hospitalization
- (7) Cranial imaging diagnosis

#### 1) NIHSS

The descriptive statistics will be calculated for the NIHSS scores at Day 4, Day 10, Day 14, after 3 weeks, at discharge, and after 3 months. The number and percentage of patients with an improvement of 4 or more points in the NIHSS score will be summarized by treatment group and analysis visit.

#### 2) mRS

The number and percentage of patients with mRS each score (0, 1,...,6) after 3 weeks, at discharge, and after 3 months will be summarized by treatment group.

#### 3) BI

The descriptive statistics for each treatment group will be calculated for the total BI score (0 to 100) at Day 14, after 3 weeks, at discharge, and after 3 months. The number and percentage of patients for BI three categorical score (100-95, 90-55, 50-0) will be summarized by treatment group and analysis visit.

#### 4) FIM

The descriptive statistics for each treatment group will be calculated for the FIM total scores (18 to 126 points) measured after 3 weeks, at discharge, and after 3 months.

The descriptive statistics will also be calculated for the motor item (13 to 91 points) and cognitive item (5 to 35 points) scores.

#### 5) Time of rehabilitation initiation

The descriptive statistics for each treatment group will be calculated for the time of rehabilitation initiation (the start date of rehabilitation minus the start date of hospitalization + 1).

#### 6) Duration of hospitalization

The descriptive statistics for each treatment group will be calculated for the duration of hospitalization (the start date of discharge minus the start date of hospitalization + 1).

(7) Cranial imaging diagnosis

#### Image analysis

#### (i) Infarct volume

The descriptive statistics for each treatment group will be calculated for the infarct volume.

# (ii) Severity of cerebral edema

The change in the edema will be calculated, and descriptive statistics for each treatment group will be calculated.

#### (iii) Presence or absence of intracranial bleeding

The proportion of subjects with intracranial bleeding will be calculated by severity, and the descriptive statistics for each treatment group will be calculated.

#### 7.2.4 Other Efficacy

Not applicable in this study.

#### 7.2.5 Quality of Life Assessments

Not applicable in this study.

| Author: | Date: 19 July, 2018 |
|---------|---------------------|

#### 7.2.6 Exploratory endpoint

#### 7.3 Safety Assessments

#### 7.3.1 Adverse Events

**Summaries** 

All AEs for each subject, including multiple occurrences of the same event, will be presented in full in a comprehensive listing including subject number, treatment, severity, seriousness, action taken, outcome, relationship to treatment, onset/stop date and duration.

AEs which start on or after dosing that are expressed or exacerbated are defined as treatment emergent adverse events (TEAEs).

The frequency and incidence of TEAEs will be summarized by System Organ Class (SOC) and Preferred Term (PT). The summary will be sorted by International Agreed Order (IAO) for SOC and alphabetical order for PT (or by frequency from the highest to the lowest).

Proportion of subjects with any TEAE, subjects with any related TEAE, subjects with any serious TEAE, and subjects with any TEAE leading to discontinuation of the study will be summarized.

Following summaries of TEAEs will be presented:

| | Summary of AEs by SOC and PT |
|---|-----------------------------------|
| П | Summary of related AEs by SOC, PT |

For summaries of AEs multiple occurrences of the same event within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the same event within a subject will be counted once in the maximum intensity category (severe > moderate > mild) and/or maximum drug relationship category (reasonable possibility>no reasonable possibility). If intensity or relationship is found to be missing the most severe occurrence will be imputed for that particular summary.

# 7.3.2 Laboratory Tests

Laboratory parameter values and changes from baseline, except for urinalysis will be summarized descriptively by analysis visit.

Clinical significance of laboratory findings will be evaluated by the Investigator with respect to pre-defined clinically relevant ranges taking into account the Investigator site's normal ranges. The laboratory data will be listed in full with clinically relevant values flagged (L=Lower than normal range, H=Higher than normal range or A=Abnormal if no reference range). A listing of laboratory values will be provided for subjects with any clinical significant findings (list relevant laboratory parameters only).

Lab parameter values and changes from baseline will be summarized descriptively by treatment group and analysis visit.

Shift tables will present the changes in clinically relevant categories from baseline to each analysis visit. The categories will be qualitative values for Urinalysis.

The test parameters(from central laboratory) are listed below.

- \* Hematology tests: White blood cell count (WBC), red blood cell count (RBC), hematocrit (Ht), hemoglobin (Hb), platelets (Plt)
- \* Blood biochemistry tests: AST (GOT), ALT (GPT), LDH, ALP, γ-GTP, total bilirubin (T-Bil), direct bilirubin (D-Bil), total cholesterol (T-Cho), triglycerides (TG), total protein (TP), CK (CPK), blood urea nitrogen (BUN), serum creatinine (Cre), eGFR, uric acid (UA), Na, K, Cl, albumin, glucose
- \* Urinalysis (qualitative): Glucose, protein, occult blood

#### 7.3.3 Vital Signs

All vital sign data will be listed.

Vital signs (systolic blood pressure, diastolic blood pressure, pulse rate, body temperature) values and changes from baseline will be summarized descriptively by analysis visit.

#### 7.3.4 12-lead ECG

All 12-lead ECG (heart rate, RR, PR, QRS, QT, QTcF, overall evaluation) parameters and findings will be listed.

12-lead ECG parameter values and changes from baseline will be summarized descriptively by analysis visit.

For ECGs, number and percentage of subjects meeting the criteria listed below will be presented:

- · QTcF > 500 msec at timepoint
- · 500≥QTcF >480msec at time point
- · 480≥QTcF >450msec at time point
- · Change from baseline in QTcF > 30 msec
- · Change from baseline in QTcF > 60 msec

Number of normal or abnormal values will be summarized by analysis visit window.

#### 7.3.5 Physical Examinations

Not applicable in the study.

#### 7.3.6 Other Safety Assessments

Neurologic Examination data will be listed.

#### 8. CHANGES FROM THE PROTOCOL

MTPC has decided that this study is prematurely terminated due to reconsideration of the MTPC's product pipeline. Therefore, the stasistical analysis plan is changed form the protocol as follows.

- Per protocol set will be excluded from the analysis populations.
- Efficacy endpoints will be only descriptively summarized without any formal statististical test.

#### 9. REVISION HISTORY FOR SAP AMENDMENTS

Version 02.00 (19 July, 2018)

• It reflects the results of the data review meeting on 18 July 2018.

# 10. DATA NOT SUMMARISED OR PRESENTED

Not applicable in the study.

#### 11. REFERENCES

# 12. VALIDATIONS

All statistical analyses will be performed using SAS version 9.3 or higher. The quality of statistical results will be ensured by double programming at Takumi Information Technology Inc.,.

#### 13. PROGRAMMING AND DATA PRESENTATION CONVENTIONS

The following sections detail all listings, tables, figures that will be produced in conjunction with the report.

For outputs, treatment groups will be represented as follows and in that order:

| Treatment Group | For Listings, Tables and Graphs |
|-------------------------------------|---------------------------------|
| Continuous infusion high-dose group | L group |
| Continuous infusion low-dose group | H group |
| Approved dosing regimen group | Control Group |

<sup>(1)</sup> Only shown where appropriate.

Listings will be presented in treatment, subject, visit (where applicable) and date (where applicable) order. Listings will be produced (landscape in MS Word) using PROC REPORT in SAS monospace font and pitch 8.

Summary tabulations will be presented by treatment group (and overall if appropriate), scheduled visit order (if appropriate). Continuous data summaries will present (unless stated otherwise) number of observations, number of missing observations (if there are any), mean, standard deviation, median, minimum and maximum. Categorical data summaries will present the number of observations and the corresponding percentage.

Number of decimal places (DP) or significant digits (SD):

Describe here the requirements, preferably in a table format, see example below:

| Statistic | Specification | Apply to |
|---|---|---|
| Minimum,<br>maximum | same number of DPs as the data provided in the datasets | All original, i.e.<br>non-derived, data<br>provided in the<br>datasets |
| mean, median, SD, confidence intervals | one more DP than<br>the raw data | All |
| Percentages | 1 DP | All |
| p-values | 3 DP | All |

#### Example guidelines for presentation of data

- Column headers in mixed case, with "(N=nn)" below treatments to denote the denominator
- decimal places aligned
- N (%) as a separate column rather than included in brackets for each element of the table,
- Categories (i.e. in column 1) in sentence case, in the order on the CRF
- Ordering of statistics N, Missing, Mean, SD, Minimum, Median and Maximum (and labelled as such). CV%, geometric means and 95% CIs for geometric mean also for PK parameters.
- Tables will be produced in landscape in MS Word using PROC REPORT in SAS monospace font and pitch 8.

# 14. LIST OF LISTINGS, TABLES AND FIGURES

The tables, figures and listings listed in this section are the minimum requirement. A complete list should be included in the SAP.

# 14.1 Listings

| No. | Title of listing | Analysis<br>Population/Dataset |
|---|---|---|
| 16.2.1 – SUBJECT DISPOSITION | | |
| 16.2.1.1 | Randomisation details | All Subjects |
| 16.2.1.2 | Subject Dispositions | All Subjects |
| 16.2.2 – ANALYSIS POPULATIONS | | |
| 16.2.2.1 | Analysis Population | All Subjects |
| 16.2.3 – DEMOGRAPHY AND BASELINE CHARACTERISTICS | | |
| 16.2.3.1 | Demography or Baseline Characteristics | All Subjects |
| 16.2.3.2 | Medical History | All Subjects |
| 16.2.3.3 | Concomitant Medications | All Subjects |
| 16.2.3.4 | Concomitant Therapys | All Subjects |
| 16.2.4 – EXPOSURE AND COMPLIANCE | | |
| 16.2.4.1 | IMP Exposure for Continuous Infusion Dosing Regimen | All Subjects |
| 16.2.4.2 | IMP Exposure for Approvel Dosing Regimen | All Subjects |
| | 16.2.5 – EFFICACY | |
| 16.2.5.1 | NIHSS | FAS |
| 16.2.5.2 | mRS | FAS |
| 16.2.5.3 | BI | FAS |
| 16.2.5.4 | FIM | FAS |
| 16.2.5.5 | Head Image Diagnosis | FAS |
| 16.2.6 – ADVERSE EVENTS | | |
| 16.2.6.1 | Adverse Events | SAF |
| 16.2.7 – OTHER SAFETY ASSESSMENTS | | |
| 16.2.7.1 | Neurological Examination | SAF |
| 16.2.7.2 | 12-lead ECG | SAF |
| 16.2.8 – | | |
| 16.2.8.1 | | All Subjects |

# 14.2 Tables

| No. | Title of table 14.1 – STUDY | Analysis<br>Population/Dataset |
|---|---|---|
| 14.1.1.1 | Analysis Populations | All Subjects |
| 14.1.1.2 | Subject Dispositions | All Subjects |
| 14.1.2.1 | Baseline Demographics | All Subjects |
| 14.1.2.2 | Medical History | All subjects |
| 14.1.2.3 | Summary of IMP Exposure for Continuous Infusion Dosing Regimen | All subjects |
| 14.1.2.4 | Summary of IMP Exposure for Approved dosing regimen | All subjects |
| | 14.2 – EFFICACY | |
| 14.2.1.1 | Summary of NIHSS (Change from Pre-NIHSS Score $\geq 4$ ) | FAS |
| 14.2.1.2 | Summary of NIHSS | FAS |
| 14.2.1.3 | Summary of mRS | FAS |
| 14.2.1.4 | Summary of BI | FAS |
| 14.2.1.5 | Summary of BI(100-95, 90-55, 50) | FAS |
| 14.2.1.6 | Summary of FIM | FAS |
| 14.2.1.7 | Summary of FIM(moter item, cognitive item) | FAS |
| 14.2.1.8 | Summary of Duration of hospatalization | FAS |
| 14.2.1.9 | Summary of Start of rehabilitation | FAS |
| 14.3 – SAFETY | | |
| 14.3.1.1 | Overall Summary of Treatment Emergent Adverse Events | SAF |
| 14.3.1.2 | Summary of Treatment Emergent Adverse Events by SAF | |
| | System Organ Class and Preferred Term | 1 |
| 14.3.1.3 | Summary of Adverse Drug Reaction by System Organ | SAF |
| ļ | Class and Preferred Term | |
| 14.3.2.1 | Summary of Hematolog | SAF |
| 14.3.2.2 | Summary of Biochemical | SAF |
| 14.3.2.3 | Summary of Urianalysis | SAF |
| 14.3.2.4 | Shift Table for Hematology | SAF |
| 14.3.2.5 | Shift Table for Biochemical | SAF |
| 14.3.2.6 | Shift Table for Urianalysis | SAF |
| 14.3.3.1 | Summary of Vital Signs | SAF |
| 14.3.4.1 | Summary of 12 lead ECG parameters | SAF |
| 14.3.4.2 | Number of Subject Meeting QTcF Criteria in 12-lead ECG | SAF |
| 14.3.4.3 | Summary of 12-lead ECG - Number of Normal/Abnomal values | SAF |
| | 14.4 – | |
| 14.4.1.1 | Summaey of | All subjects |

#### 15. APPENDIX 1 – ANALYSIS TIME WINDOW

#### Data handling (Safety and Efficacy assessment)

The acceptable windows of the visit of evaluations and measurements are as follows:

| Period | Visit | Targeted<br>Study<br>Days* | Analysis Visit | Analysis Visit Window in<br>Study Days |
|---|---|---|---|---|
| Befor<br>Treatment<br>Initiation | Confirmation of suitability | 0 | Baseline | [0, 1 (Day 1 prior to treatment initiaion)] ** |
| Study Drug<br>Treatment | Day 1 | 1 | Day 1 | 1 (Day 1 after treatment initiation) |
| Period | Day 2 | 2 | Day 2 | 2 |
| | Day 3 | 3 | Day 3 | 3 |
| | Day 4 | 4 | Day 4 | 4 or [3, 4]*** or [4, 6]*** |
| | Day 5 | 5 | Day 5 | 5 |
| | Day 7 | 7 | Day 7 | [6, 8] |
| 1 | Day 10 | 10 | Day 10 | [9, 11] |
| | Day 14 | 14 | Day 14 | [14, 15] |
| | Study drug | _ | Study drug | [Study drug treatment |
| | treatment period | | treatment | period discontinuation day, |
| | discontinuation | | period discontinuation | Study drug treatment period discontinuation day + 1] |
| Observation | After 3 weeks | 22 | After 3 weeks | [20, 24] |
| period | At discharge | - | At discharge | [At discharge day - 1, At discharge day] |
| | After 3 months or<br>at observation<br>period<br>discontinuation | 85 | After 3 months | [77, 93] |
| | At observation period discontinuation | - | At observation period discontinuation | [At observation period discontinuation day, At observation period discontinuation day +8] |

<sup>\*</sup> Study days will be calculated from the first dose of study drug.

<sup>\*\*</sup> The neurological assessments at baseline will be performed once in the period from the time of consent acquisition to Day 5.

<sup>\*\*\*</sup> Labolatory tests, Vital signs and 12-Lead ECG will be measured before continuous intravenous injection of 72 hours (-1 day) and Head Image Diagnosis will be taken after continuous intravenous injection of 72 hours (2 days).